CLINICAL TRIAL: NCT03877692
Title: Acute Control of Chronic Hypertension in Preeclampsia
Brief Title: Acute Control of Chronic Hypertension
Acronym: ACCTIVE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5253
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Preeclampsia With Severe Features; Chronic Hypertension in Obstetric Context
Keywords: Hypertension; Labetalol
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principle investigator and outcomes assessor are masked to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental labetalol dose (Experimental): Subjects receive 40mg, 60mg, 80mg after each severe BP
  Interventions: Drug: Experimental dosing of labetalol
- Current standard of care (Active Comparator): Subjects receive 20mg, 40mg, 60mg after each severe BP
  Interventions: Other: Standard dosing of labetalol

INTERVENTIONS:
Drug: Experimental dosing of labetalol — Subjects with preexisting hypertension who have sustained severe hypertension (SBP≥160 mmHg and/or DBP≥110 mmHg), 15 min apart receive the experimental dosing of labetolol. Subjects in both groups are managed following the standard guidelines established by ACOG (Committee Opinion #623). For each successive episode of hypertension treatment, patients are asked a set of questions to monitor for adverse medication side-effects. The fetus is electronically monitored for four hours after the last IV dose.
  Arms: Experimental labetalol dose
Other: Standard dosing of labetalol — Subjects with preexisting hypertension who have sustained severe hypertension (SBP≥160 mmHg and/or DBP≥110 mmHg), 15 min apart receive either the standard of care dosing of labetolol. Subjects in both groups are managed following the standard guidelines established by ACOG (Committee Opinion #623). For each successive episode of hypertension treatment, patients are asked a set of questions to monitor for adverse medication side-effects. The fetus is electronically monitored for four hours after the last IV dose.
  Arms: Current standard of care

SUMMARY:
The purpose of this study is to understand if administration of a personalized dose of the anti-hypertensive medication, labetalol, based on patient's history of preexisting hypertension, will be more effective at controlling severe hypertension during pregnancy, compared to the current standard dosing.

DETAILED DESCRIPTION:
The investigators seek to asses the effect of preexisting hypertension on the patient's response to treatment for severe hypertension in preeclampsia with severe features. The investigators hypothesize that successive administration of 40-60-80 mg of labetolol will reduce time to blood pressure control versus the standard dosing, 20-40-80 mg labetolol, recommended by the American College of Obstetricians and Gynecologists in 2015.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Gestational age ≥ 24 weeks
* Singleton gestation
* Chronic hypertension as defined as two elevated blood pressures (SBP ≥ 140mmHg and/or DBP ≥ 90mmHg) at least 4 hours apart before 20 weeks gestation

Exclusion Criteria:

* Known allergic reaction to labetalol
* Persistent mild-moderate asthma (≥ 2 rescue inhaler uses per week in the previous month)
* Obstructive airway disease
* Bradycardia < 70 beats/min
* Heart block > 1st degree or history of heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Time to blood pressure control | This outcome will be measured during antepartum admission and will start with the first dose of IV labetalol given for severe blood pressure until subsequent blood pressure check is non-severe (<160 systolic and <110 diastolic), ending with delivery
  length of time in minutes between IV labetalol treatment and non-severe blood pressure
Length of blood pressure control | This outcome will be measured during antepartum admission and will start with the first non-severe blood pressure after IV labetalol dosing until the next dose of IV labetalol is indicated (by severe blood pressure), ending with delivery
  length of time in minutes between successful treatment resulting in non-severe blood pressure and need for next dose of IV labetalol

SECONDARY OUTCOMES:
Maternal adverse events | within 3 months of delivery
  Anticipated and unanticipated adverse events experienced by the mother including Symptomatic hypotension, bradsycardia, bronchospam, seizure, stroke, death
Neonatal adverse events | within 28 days of delivery
  Any complications experienced by the neonate including APGAR score < 5, need for respiratory support, blood glucose, death

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Obstetrics and Gynecology, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee Opinion No. 623: Emergent therapy for acute-onset, severe hypertension during pregnancy and the postpartum period. Obstet Gynecol. 2015 Feb;125(2):521-525. doi: 10.1097/01.AOG.0000460762.59152.d7. PMID 25611642